CLINICAL TRIAL: NCT02423096
Title: Neuroendocrine, Metabolite Substrates, Clinical Symptoms and Cognitive Function in Schizophrenia
Brief Title: Neuroendocrine and Metabolite Substrates in Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang Liang-Jen, Associate Professor and Visiting Staff, Chang Gung Memorial Hospital
Other Study IDs: 103-0721C
Record Dates: First submitted 2015-04-15; First posted 2015-04-22 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
Keywords: biomarker; neuroendocrine; metabolite; cognitive functioning; clinical symptoms; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Haloperidol; Sulpiride; Olanzapine; Quetiapine Fumarate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Biospecimen Retention: Samples Without DNA — Blood samples of patients and control subjects will be obtained to measure the levels of neuroendocrine substrates (didehydroepiandrosterone, dehydroepiandrosterone sulfate, pregnenolone, and cortisol) and metabolite markers (lipid profiles, glycerate, eicosenoic acid, pyruvate, b-hydroxybutyrate, Cysteine)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Schizophrenia: Patients with schizophrenia will be treated with antipsychotic drugs as routine care (i.e., risperidone, haloperidol, sulpiride, olanzapine, quetiapine).
  Interventions: Drug: Risperidone
- Healthy controls: No special intervention will be provided for healthy controls.

INTERVENTIONS:
Drug: Risperidone — Patients with schizophrenia will be treated with antipsychotic drugs as routine care.
  Other Names: Haloperidol; Sulpiride; Olanzapine; Quetiapine
  Groups: Schizophrenia

SUMMARY:
Background: Schizophrenia is a serious mental illness. The diagnosis and severity evaluations of schizophrenia are generally based on patient behaviors. Biomarkers are objectively measured and used as indicators for diagnosis confirmation, symptom assessment, and evaluation of pharmacologic responses to therapeutic interventions. Neuroendocrine and metabolite substrates are potential biomarkers of the pathogenic processes in schizophrenia.

Aims: The aims of this study are to determine (a) the differences in neuroendocrine and metabolite substrates between patients diagnosed with schizophrenia and healthy controls; and (b) the associations among the neuroendocrine and metabolite substrates, cognitive function, clinical symptoms, and treatment responses of patients diagnosed with schizophrenia.

Methods: (a) The investigators plan to recruit 100 patients diagnosed with schizophrenia and 100 healthy controls as participants. (b) At the baseline and Week 12, patient blood samples will be obtained to measure the levels of neuroendocrine substrates and metabolite markers. Clinical symptoms and cognitive function will be evaluated. (c) For the healthy control participants, blood samples will be obtained once to measure neuroendocrine and metabolite marker levels.

Expected Results: The results of this study may contribute to identifying potential neuroendocrine and metabolite biomarkers of schizophrenia, and clarify the associations among the neuroendocrine and metabolite substrates, cognitive function, clinical symptoms, and treatment responses of patients diagnosed with schizophrenia. Such information is crucial for clinical evaluations and future research.

DETAILED DESCRIPTION:
1. The investigators plan to recruit 100 patients with schizophrenia and 100 healthy control subjects.
2. For the patients, diagnoses of schizophrenia will be confirmed using the Chinese version of the Mini International Neuropsychiatric Interview (MINI). At the baseline and Week 12, patient blood samples will be obtained to measure the levels of neuroendocrine substrates (didehydroepiandrosterone, dehydroepiandrosterone sulfate, pregnenolone, and cortisol) and metabolite markers (lipid profiles, glycerate, eicosenoic acid, pyruvate, b-hydroxybutyrate, Cysteine). Cognitive function will be evaluated using the Brief Assessment of Cognition in Schizophrenia. The participants' clinical symptoms and daily activities will be assessed using the Positive and Negative Syndrome Scale, 17-item Hamilton Depression Rating Scale, and Personal and Social Performance Scale.
3. For the healthy control subjects, psychiatric diagnoses will be verified using MINI, and blood samples will be obtained once to measure neuroendocrine and metabolite marker levels.

ELIGIBILITY:
Patients with Schizophrenia

Inclusion criteria:

1. Diagnosed with schizophrenia and will be confirmed using the Chinese version of the Mini International Neuropsychiatric Interview (MINI).
2. Age between 18 to 79.
3. Have signed the informed consent.

Exclusion criteria:

1. Having history of illicit drug use or other major psychiatric disorders (e.g., bipolar disorder, major depressive disorder, or organic mental disorders).

Healthy Controls

Inclusion criteria:

1. Psychiatric diagnosis without schizophrenia will be confirmed using the Chinese version of MINI.
2. Age between 18 to 79.
3. Have signed the informed consent.

Exclusion criteria:

1. Having history of illicit drug use or other major psychiatric disorders (e.g., psychosis, bipolar disorder, major depressive disorder, or organic mental disorders).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients with schizophrenia will be recruited from the out-patient department in Kaohsiung Chang Gung Memorial Hospital, Kaohsiung city, Taiwan
  2. Healthy controls will be recruited from the staff in Kaohsiung Chang Gung Memorial Hospital and from the communities in Kaohsiung city, Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale | Participants will be assessed at the outpatient department, an expected average of 30 min.

SECONDARY OUTCOMES:
Brief Assessment of Cognition in Schizophrenia | Participants will be assessed at the outpatient department, an expected average of 40 min.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Jen Wang, MD, MPH, Principal Investigator — Chang Gung Memorial Hospital, Kaohsiung, Taiwan
Locations (1):
- Liang-Jen Wang, Kaohsiung City, Kaohsiung, Taiwan